CLINICAL TRIAL: NCT04484506
Title: A Prospective Phase II Study of Pegaspargase-COEP Chemotherapy Combined With Radiotherapy for Patients With Newly Diagnosed Extra-nodal NK/T-cell Lymphoma
Brief Title: Pegaspargase-COEP Chemotherapy Combined With Radiotherapy for Extra-nodal NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Peking University International Hospital (Other); Hebei Medical University Fourth Hospital (Other); Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhu, Dr., Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COEPL for NKTCL
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: NK/T Cell Lymphoma Nos
MeSH Terms: interventions — pegaspargase; Cyclophosphamide; Vincristine; Etoposide; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage I/II nasal ENKTL (Experimental): 2-3 cycles of induction pegaspargase-COEP chemotherapy followed by concurrent chemoradiotherapy, then by 1-2 cycles of pegaspargase-COEP chemotherapy as consolidation
  Interventions: Drug: pegaspargase, cyclophosphamide, vincristine, etoposide, prednisone
- Stage III/IV or primary extra-nasal ENKTL (Experimental): 6-8 cycles of pegaspargase-COEP chemotherapy with or without local radiotherapy and/or consolidative autologous stem cell transplantation
  Interventions: Drug: pegaspargase, cyclophosphamide, vincristine, etoposide, prednisone

INTERVENTIONS:
Drug: pegaspargase, cyclophosphamide, vincristine, etoposide, prednisone — Cyclophosphamide 750 mg/m2 intravenously on day 1, vincristine 1.4 mg/m2 intravenously on day1, etoposide 60mg/m2 intravenously on days 1-3; pegaspargase 2500IU/m2 intramuscularly on day 2, prednisone 100mg orally on days 1-5.

SUMMARY:
The optimal first-line treatment for extra-nodal NK/T-cell lymphoma (ENKTL) has not been well-defined. This phase II study aimed to evaluate the efficacy and safety of pegaspargase, cyclophosphamide, vincristine, etoposide and prednisone (COEPL) regimen combined with radiotherapy for patients with newly diagnosed ENKTL.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed pathological diagnosis of ENKTL as defined by WHO criteria
* age 14-80 years
* no prior chemotherapy or radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* at least one measurable lesion
* adequate bone marrow function (i.e. hemoglobin ≥80 g/l, absolute neutrophil count ≥ 1.0 × 10^9/L, platelets ≥ 100 ×10^9/L), adequate renal function (i.e. serum creatinine ≤177 μmol/L), adequate hepatic function (e.g. total bilirubin ≤ two times the upper limit of normal, and ALT /AST ≤2.5 times the upper limit of normal)
* expected survival of more than three months

Exclusion Criteria:

* invasion of lymphoma to central nervous system
* pre-existing coagulation disorder
* other concomitant neoplasms
* severe infection
* positive HIV antibody
* HBV DNA titer higher than 10^4 copies /ml in HBsAg-positive patients post antiviral therapy
* pregnant or lactating women
* women of childbearing age unwilling to take contraceptive measures during the study period

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-10-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 1 year

SECONDARY OUTCOMES:
Overall response rate | 1 year
Progression-free survival | 3-year
Overall survival | 3-year
Adverse events | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No